CLINICAL TRIAL: NCT06975670
Title: ENHANCING COMPREHENSION OF INFORMED CONSENT IN RESEARCH INVOLVING PATIENTS WITH PSYCHOTIC DISORDERS USING AUDIO-VISUAL AIDS
Brief Title: Enhancing Comprehension of Consent in Patients With Psychotic Disorders
Acronym: UBACC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Makerere University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: Mak-SOMREC-2022-478; GRANT NUMBER D43TW010892) (Other Grant/Funding Number: NIH)
Record Dates: First submitted 2025-05-09; First posted 2025-05-16 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Psychosis
MeSH Terms: conditions — Psychotic Disorders

STUDY DESIGN:
Intervention Model Description: To randomize participants into two consent arms. The control arm are those who will be given routine traditional paper consent, then the intervention arm, those who will be given a multimedia consent tool and assess if their is improvement in comprehension
Who Masked: Investigator, Outcomes Assessor
Masking Description: They will not know the arm that the patient belonged to during asssesment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention arm (Other): The 30 participants assigned to the multimedia consent, which is the intervention arm, will first meet individually with a trained research assistant who will provide a video that explains the protocol and encourage them to watch it. Subjects will be encouraged to have the RA stop the multimedia consent video and repeat any segments that are unclear. Participants will also be encouraged to discuss and clarify issues with the RAs (and not simply have the video rerun). Having such a discussion is vital in that, much as multimedia consent aids appear to be more effective as aids, they should not be viewed as substitutes for person-to-person interaction(Flory & Emanuel, 2004). In order to control for social element consent enhancement, the role of the RA will be emphasized that he or she is meant to guide the participant, not educating them. The RA will record duration of time the consent will takes for each participant, so that we compare time spent in each consent condition.
  Interventions: Other: multimedia consent tool
- control arm (No Intervention): The 30 participants assigned to the routine paper consent procedure which is the control arm, will first meet individually with a trained research assistant who will provide the subjects with the printed consent form and encourage them to read along while the research assistant (RA) read it aloud. Participants will be motivated to stop the RA and seek for clarification any time during the consent process. To control for social element consent enhancement, the role of the RA will be emphasized that he or she is meant to guide the participant, not educating them. The RA will record duration of time the consent will take for each participant, so that we compare time spent in each consent condition

INTERVENTIONS:
Other: multimedia consent tool — The multimedia consent tool is new and developed for this particular study
  Arms: Intervention arm

SUMMARY:
: Informed consent is an important aspect of research, however in psychiatry research it remains an ethical dilemma, for the lack of clarity on the consent process deters some researchers from mental health research, and yet a good research must ensure that this moral stand is undertaken. Studies that literally test measures that improve the informed consent process in participants with psychotic disorders have been scanty. To date, there is a noticeable absence of an evidence-based intervention for enhancing the comprehension of consent information in research participants with psychotic disorders in the Ugandan context. Thus, this research study is to explore methods like incorporating multimedia components, such as audio and visual aids, to enhance the participants' grasp of research particulars, thereby enabling them to make informed decisions effectively and give informed consent when they are invited to participate in research projects.

Objective: To evaluate the comprehension of informed consent, identify key factors that that are associated with comprehension of consent, and determine the feasibility, acceptability, and preliminary effectiveness of audio-visual aids on enhancing the comprehension of consent information during the consenting process in research involving individuals with psychotic disorders.

Methods: This will be a multi-method research design that will be achieved through four sub-studies. Sub-study 1 will be cross-sectional and will involve an assessment of comprehension of informed consent using the University of California Brief Assessment of Capacity to Consent (UBACC) tool. Participants will be patients aged 18- 60 years with a psychotic disorder. Sub-study 2 will be a qualitative study that utilizes a user-centered design approach by engaging a multidisciplinary team of stakeholders to develop a multimedia audio-visual consent tool.

Sub-study 3 will be a randomized pilot study designed to evaluate the effectiveness of the multimedia video consent tool and how it compares with the traditional paper method in enhancing participants' comprehension of consent information.

Sub-study 4 will be a mixed-methods approach using quantitative and qualitative data from exit interviews to assess the Feasibility and Acceptability of the audio-visual consent tool for individuals with psychotic disorders and the research assistants administering the tool in a mental health research setting

DETAILED DESCRIPTION:
Scope of the Study Depth of Investigation

The study aims to evaluate the comprehension of informed consent among participants with psychotic disorders using quantitative methods. It is also set to develop and evaluate the effectiveness of audio-visual aids in enhancing comprehension of consent research information compared to traditional paper-based consent methods using both qualitative and quantitative methods. The investigation involves:

1. Quantitative Analysis: Assessing comprehension levels using the University of California, San Diego Brief Assessment of Capacity to Consent (UBACC) tool.
2. Qualitative Analysis: Developing and pilot-testing a multimedia audio-visual consent tool through stakeholder consultations.
3. Comparative Analysis: Conducting a randomized pilot study to compare the effectiveness of routine paper consent with multimedia audio-visual consent.

Content The study content encompasses the development of a multimedia audio-visual consent tool, informed by input from a multidisciplinary team, including mental health professionals, ethicists, Information technologists and participants' representatives. It involves the application of multi-method research design, integrating both descriptive and thematic analyses, as well as statistical evaluations using logistic regression and mixed-effects linear regression models.

Sample Size The study will involve participants diagnosed with psychotic disorders who are engaged in mental health services in Butabika National Referral Psychiatric Hospital in Uganda, hereafter referred to as Butabika Hospital A representative sample size will be determined based on power calculations to ensure the reliability and validity of the findings.

Geographical Coverage The research will be conducted in Uganda, specifically focusing on in-patients and outpatients with a psychotic disorder at Butabika Hospital who will be present during the study period and fulfill the selection criteria. This geographical focus allows for an examination of context-specific challenges and opportunities in the consent process.

Time Frame The study is designed to be conducted over a period of two years, allowing for comprehensive data collection, tool development, pilot testing, and analysis. This time frame ensures thorough investigation and iterative refinement of the consent process and materials.

Theoretical Coverage The study is grounded on the cognitive theory of multimedia learning and dual coding together with ethical principle that emphasize autonomy and informed consent in mental health research. It draws on these theories to explore how multimedia tools can enhance comprehension, thus decision-making among participants with psychotic disorders.

ELIGIBILITY:
Inclusion Criteria:

* Psychotic disorders who score below 14.5 on UBACC trials.
* 18-60 years

Exclusion Criteria:

* Those participants that do not speak English or Luganda will be excluded from the study
* Hearing or Visual impairments

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05-30 (Estimated); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Enhanced comprehension of consent information | 1 week
  Shall use the measure of the scores for the UBACC tool

CONTACTS AND LOCATIONS:
Overall Officials: Ponsiano Ochama, PhD, Study Chair — Makerere University

IPD SHARING:
Plan to Share IPD: Yes
Data will be deposited in the repository,
Supporting Information: Study Protocol, SAP, ICF
Time Frame: As advised